CLINICAL TRIAL: NCT02201121
Title: Influences of Phenylephrine, Dopamine and Ephedrine on Stroke Volume Variation and Pulse Pressure Variation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ran Kong, Department of Anesthesiology, People's Liberation Army General Hospital, Beijing, China, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: plaghran001
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2013-10

CONDITIONS: Circulation; Drug Dose; Calculated SAP
MeSH Terms: interventions — Dopamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- phenylephrine group, dopamine group, ephedrine group (Experimental): phenylephrine group: use the phenylephrine to increase the SAP from low to high level.
  dopamine group: use the dopamine to increase the SAP from low to high level. ephedrine group:use the ephedrine to increase the SAP from low to high level.
  Interventions: Other: Influences of phenylephrine, dopamine and ephedrine on stroke volume variation and pulse pressure variation

INTERVENTIONS:
Other: Influences of phenylephrine, dopamine and ephedrine on stroke volume variation and pulse pressure variation — This research mainly study the effect of clinical commonly used vasoconstrictor drugs on blood pressure of pressure

SUMMARY:
Although induced hypertension decreased SVV and PPV,the influences of stroke volume variation and pulse pressure variation caused by phenylephrine,dopamine and ephedrine were unknown.

DETAILED DESCRIPTION:
Pulse pressure variation (PPV) and stroke volume variation (SVV) during mechanical ventilation have been shown to be effective parameters to predict preload responsiveness. Although induced hypertension decreases PPV and SVV, the influences of phenylephrine, dopamine and ephedrine on PPV and SVV are unknown.

ELIGIBILITY:
Inclusion Criteria:

* Their American Society of Anesthesiologists (ASA) physical status was 1 or 2
* Body mass index (BMI) ranged from 18 to 26
* None of the patients had known diabetes mellitus, hypertension, cardiovascular, pulmonary, endocrinological, neurological diseases, or diseases that influenced intravascular fluid volume or balance
* All patients had a preoperative fast for at least 8 h and routine atropine intramuscular injection

Exclusion Criteria:

* Persistent arrhythmias
* Intraoperative application of vasoactive drugs except phenylephrine, dopamine and ephedrine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
invasive arterial blood pressure as a Measure of Safety | DAY 1
  if instability of circulation, stop the clinical trial